CLINICAL TRIAL: NCT06466603
Title: A Randomized, Double-blind, Placebo-controlled Study with Open-Label Extension Investigating the Effects of 2 Different Doses of GABA Probiotic Lp815 on Anxiety in Individuals with Mild to Moderate Anxiety in a Home Setting
Brief Title: Probiotics for Anxiety Study
Status: Active, not recruiting | Type: Observational
Sponsor: Verb Biotics LLC (Industry)
Collaborators: People Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PS08
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Anxiety
Keywords: Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- GABA Probiotic Dose 1: Dose 1 is a GABA Probiotic containing Lactiplantibacillus plantarum 815 (1 Billion cfu/dose). Capsule taken once daily with food.
  Interventions: Dietary Supplement: GABA Probiotic Dose 1
- GABA Probiotic Dose 2: Dose 2 is a GABA Probiotic containing Lactiplantibacillus plantarum 815 (5 Billion cfu/dose).
  Capsule taken once daily with food.
  Interventions: Dietary Supplement: GABA Probiotic Dose 2
- Placebo Group: Non-active ingredients in the probiotic capsule include organic rice maltodextrin. Capsule taken once daily with food.
  Interventions: Dietary Supplement: Placebo Group

INTERVENTIONS:
Dietary Supplement: GABA Probiotic Dose 1 — Participants will complete up to a seven week study consisting of screening period, baseline period, up to a 6-week product use period with a total of 42 product use sessions. Screening assessments, baseline questions, product use period questionnaires, adverse event reporting, and end of study experience survey data will be collected. After the 6-week study product use period, all participants will be given the option to continue using GABA Probiotic for an additional 4 weeks. This study will be conducted remotely and will use a web-based data collection platform, Consumer Health Learning and Organizing Ecosystem (Chloe), by People Science where participants will complete study assessments using the Chloe app during the course of the study. Participants will receive the study product during the baseline period. Demographic and medical history data will be collected for the study.
  Groups: GABA Probiotic Dose 1
Dietary Supplement: GABA Probiotic Dose 2 — Participants will complete up to a seven week study consisting of screening period, baseline period, up to a 6-week product use period with a total of 42 product use sessions. Screening assessments, baseline questions, product use period questionnaires, adverse event reporting, and end of study experience survey data will be collected. After the 6-week study product use period, all participants will be given the option to continue using GABA Probiotic for an additional 4 weeks. This study will be conducted remotely and will use a web-based data collection platform, Consumer Health Learning and Organizing Ecosystem (Chloe), by People Science where participants will complete study assessments using the Chloe app during the course of the study. Participants will receive the study product during the baseline period. Demographic and medical history data will be collected for the study.
  Groups: GABA Probiotic Dose 2
Dietary Supplement: Placebo Group — Participants will complete up to a seven week study consisting of screening period, baseline period, up to a 6-week product use period with a total of 42 product use sessions. Screening assessments, baseline questions, product use period questionnaires, adverse event reporting, and end of study experience survey data will be collected. After the 6-week study product use period, all participants will be given the option to continue using GABA Probiotic for an additional 4 weeks. This study will be conducted remotely and will use a web-based data collection platform, Consumer Health Learning and Organizing Ecosystem (Chloe), by People Science where participants will complete study assessments using the Chloe app during the course of the study. Participants will receive the study product during the baseline period. Demographic and medical history data will be collected for the study.
  Groups: Placebo Group

SUMMARY:
The purpose of this study is to observe the effect of a consumer-grade probiotic capsule called GABA (gamma-aminobutyric acid ) Probiotic ("Study Product"), a probiotic capsule containing Lactiplantibacillus plantarum 815, on anxiety. The purpose of this study is to evaluate the effects of 2 different doses of this probiotic study product on anxiety in comparison to placebo. Additionally, the study aims to observe the effects of the probiotic study product on mood, cognitive function, quality of life and sleep. After the 6-week study product use period, all participants will be given the option to continue using GABA Probiotic for an additional 4 weeks.

Participants in this study will complete surveys and questionnaires about their experience before, during and after taking the study product. Additionally, this study will incorporate the use of a wrist-worn electronic device to measure sleep.

DETAILED DESCRIPTION:
This study aims to observe the effect of Lactiplantibacillus plantarum VDL815 formulated into a probiotic capsule in individuals with mild to moderate anxiety to serve as a pilot exploration of potential health benefits and dosing. Participants will complete up to a 16-week study consisting of a screening period, randomization and shipping period, a baseline period, a 6-week product/placebo use period and an optional 4-week open label extension.

The rationale for this study is to observe the effect of 2 different doses of a consumer-grade probiotic capsule called GABA Probiotic on anxiety in individuals with mild to moderate anxiety. Additionally, the study aims to observe the effects of the probiotic product on mood, cognition, quality of life, and sleep disturbance. A consumer-driven, decentralized observational clinical research study is well-suited for examining the effect of this probiotic on anxiety.

Anxiety is highly prevalent and impacted by many interdependent variables. We will examine self-reported anxiety in a broad age-range of adults who have chosen to try this product. The study will incorporate participant reported outcome questionnaires and surveys and the use of a health tracking wearable device to explore objective digital outcome measures of sleep and heart rate variability. There is no "doctor-patient" relationship as part of this research since the participant as a consumer is making the informed choice to take the product and take part in the observational process with self-reported measures. Findings from this study will contribute knowledge toward the dosing and formulation of the probiotic product and the design of future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Has self-reported mild to moderate generalized anxiety
* Generalized Anxiety Disorder-7 (GAD-7) score of 5-14 at screening
* Interested in understanding more about their anxiety and the use probiotic products
* If taking any OTC or other products for anxiety and/or sleep (e.g. magnesium, melatonin, anticholinergics etc.), must be on a stable dose for at least 4 weeks prior to randomization and maintain the stable intake for the duration of the study.
* Willing to do a 4-week washout from any systemic antibiotic use prior to randomization.
* If using any cannabis-containing products, must be on a stable dose for at least 4 weeks prior to randomization.
* In good general health at the time of screening (Investigator discretion).
* Able to read and understand English.
* Able to read, understand, and provide informed consent.
* Able to use a personal smartphone device and download Chloe by People Science.
* Able to receive shipment of the product at an address within the United States.
* Willing to wear a health tracking wearable device everyday (up to 7 weeks) during sleep.
* Able to complete study assessments over the course of up to 7 weeks.

Exclusion Criteria:

* Do not have a smartphone and/or internet access.
* Concomitant Therapies:

  * Participants taking prescription medication for anxiety and/or sleep
  * Participants receiving any investigational therapies or treatments within 30 days prior to randomization.
* Other Illnesses or Conditions: Participants who have the following co-morbidities are excluded:

  * Known diagnosis of Generalized Anxiety Disorder that is uncontrolled and severe
  * Known diagnosis of Inflammatory Bowel Disease
  * Known diagnoses of the following disorders: Narcolepsy, Restless Leg Syndrome, Circadian Rhythm Disorders, Panic Disorder
  * Current or prior psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample size for this study will be approximately 122 healthy volunteers who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2025-02-11 (Estimated)

PRIMARY OUTCOMES:
To observe the effect of the 2 different doses of the study product on anxiety | 7 Weeks
  Change in Generalized Anxiety Disorder-7 (GAD-7) score by 4 points between placebo and study product groups. Baseline period will be compared as well GAD-7 scores between the 2 doses. Scores range from 0 to 21, higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
To assess the effect of 2 different doses of the study product symptoms of sleep disturbance | 7 Weeks
  Change in the Insomnia Sleep Index (ISI) score by 4.5 points between placebo and study product groups. Baseline period will be compared as well ISI scores between the 2 doses. Scores range from 0 to 28, higher scores indicating a worse outcome.
To assess the effect of 2 different doses of the study product on sleep quality | 7 Weeks
  Change in average sleep quality score by 1 point as measured by daily 11-point visual analogue rating scale (VAS) between placebo and study product groups. Baseline period will be compared as well as average scores between the 2 doses. Scores range from 0 to 10, higher scores indicating a better outcome.
To assess the effect of 2 different doses of the study product on quality of life | 7 Weeks
  Change in average mood score by 1 point between placebo and study product groups as measured by a daily 5-point VAS scale. Baseline period will be compared as well the scores between the 2 doses. Scores range from 1 to 5, higher scores indicating a better outcome.
To assess the effect of 2 different doses of the study product on cognitive ability | 7 Weeks
  Change in average score between placebo and study product groups on the Cognitive Assessment: Raven's Progressive Matrices collected weekly. Baseline period will be compared as well the scores between the 2 doses. Scores range from 0 to 10, higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Craft, MD, Principal Investigator — People Science, Inc.
Locations (1):
- People Science, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grant AD, Erfe MCB, Delebecque CJ, Keller D, Zimmerman NP, Oliver PL, Youssef B, Moos J, Luna V, Craft N. Lactiplantibacillus plantarum Lp815 decreases anxiety in people with mild to moderate anxiety: a direct-to-consumer, randomised, double-blind, placebo-controlled study. Benef Microbes. 2025 Apr 24;16(5):521-532. doi: 10.1163/18762891-bja00073. PMID 40312029